CLINICAL TRIAL: NCT05064267
Title: Evaluation of Thrombelastography vs. Non-Viscoelastic Assays to Predict Hypercoagulability in Pediatric Chronic Kidney Disease: A Pilot Study
Brief Title: Hemostatic Profiles in Pediatric CKD
Status: Completed | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00000777
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Kidney Disease, Chronic; Pediatric Kidney Disease; Renal Insufficiency, Chronic; Blood Coagulation Disorders in Children
Keywords: thromboelastography; TEG; viscoelastic assay
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CKD stage 3: Between the ages of 6 months and 17 years currently followed within the hospital system's CKD clinic, and diagnosed with CKD 3 from a non-inflammatory etiology.
  Interventions: Diagnostic Test: phlebotomy
- CKD stage 4: Between the ages of 6 months and 17 years currently followed within the hospital system's CKD clinic, and diagnosed with CKD 4 from a non-inflammatory etiology.
  Interventions: Diagnostic Test: phlebotomy
- CKD stage 5: Between the ages of 6 months and 17 years currently followed within the hospital system's CKD clinic, and diagnosed with CKD 5 from a non-inflammatory etiology.
  Interventions: Diagnostic Test: phlebotomy

INTERVENTIONS:
Diagnostic Test: phlebotomy — phlebotomy will be performed to obtain coagulation labs of interest. Specifically, in addition to standard clinical labs, the following will be drawn on study participants: thrombelastography with platelet mapping, antithrombin, DIC panel, factor VIII, vWF antigen, Protein C antigen and activity, Protein S antigen and activity, and ferritin.

SUMMARY:
This cross-sectional pilot study will examine the blood clotting patterns in children with chronic kidney disease stages 3, 4, and 5. A total of 30 participants will be enrolled with 10 participants for each stage of chronic kidney disease. Blood specimens will be collected from each participant during a routine clinic visit, and will then be processed to evaluate blood clotting characteristics according to thrombelastography and more conventional clotting tests.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is associated with 5% of all pediatric inpatient venous thromboembolism (VTE) occurrences, but rates of occurrence are likely underreported in current literature. VTE is associated with a 2-fold increase in mortality, and exponentially higher rates of healthcare expenditure. Because VTE is a low-incidence but high-impact complication of CKD, evaluating those at risk presents a unique challenge. The underlying pathophysiology of thrombosis in CKD is poorly understood, but likely involves changes across the hemostatic and fibrinolytic systems. Standard laboratory tests provide a poor representation of in-vivo clot formation, particularly in the complex hemostatic environment of CKD, as these tests undergo centrifugation and much of the cellular debris known to contribute to clot formation is lost. Viscoelastic assays are a reemerging tool that provide a qualitative measure of each hemostatic milestone, from clot formation through degradation, in whole-blood; thereby preserving the cellular debris and additional factors that contribute to clot formation in-vivo.

The purpose of this study is to evaluate the utility of Thrombelastography vs conventional clotting tests to predict onset of hypercoagulability and the relationship to the stage of pediatric Chronic Kidney Disease (CKD). The investigators hypothesize that as kidney function deteriorates, a more pronounced prothrombotic profile is expected to emerge according to TEG and conventional clotting tests. This will be demonstrated by an overall increase in measured values across the coagulation portion of the TEG and a decrease in the measured fibrinolysis. According to conventional clotting tests, it is expected to find increased levels of Factor VIII antigen, Fibrinogen, vWF, Protein C/S, and D-dimer. Depending upon an individual's degree of proteinuria, levels of Antithrombin would be expected to decrease as it is lost in the urine. This urinary loss of Antithrombin would also contribute to an overall prothrombotic profile.

This cross-sectional pilot study will enroll 30 participants between the ages of 6 months and 17 years who have been previously diagnosed with CKD stages 3, 4, or 5. Enrollment will occur during a routine clinic visit wherein the participant was also previously scheduled to receive venipuncture for ongoing monitoring of labs. Study specific lab values, in addition to routine lab values of interest and pertinent past medical history, will be extracted from the EMR.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients ages 6 months - 17 years
* Currently followed in the CKD clinic at Children's Healthcare of Atlanta (CHOA)
* Diagnosed with Stage 3, Stage 4 or Stage 5 CKD
* Must have routine venous laboratory tests planned as a component of their clinic encounter.

Exclusion Criteria:

* Participants <13.6kg (to allow for safe blood sample volumes).
* History of venous thromboembolism, post solid organ transplant, co-diagnosis of inflammatory disease, and nephritis.
* Personal or family history of inherited thrombophilia conditions
* Hospital admission within the last 30 days.
* Transfusion (PRBC, FFP, Platelets, or Cryoprecipitate) within the last 30 days.
* Those on the following medications: steroids and anti-coagulants.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Previously established, and routinely followed, pediatric individuals between the ages of 6 months and 17 years with a non-inflammatory etiology of chronic kidney disease staged as 3, 4, or 5.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Degree of statistically-significant correlation between conventional clotting tests and thrombelastography when determining the degree of hypercoagulability for pediatric patients diagnosed with chronic kidney disease stages 3, 4, and 5 | Day 1
  Thrombelastography with platelet mapping, antithrombin, vwF, Factor VIII antigen, DIC panel, Protein C activity and antigen, Protein S activity and antigen, and Ferritin labs will be evaluated in each participant from the 3 CKD groups.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Calamaro, PhD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No